CLINICAL TRIAL: NCT02378701
Title: Interventional Validation of an MDS-Specific Measure of Quality of Life: Assessing the Responsiveness of the Quality of Life in Myelodysplasia Scale (QUALMS-1) to Different Hypomethylating Agent Regimens for Low and Intermediate Risk Disease
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: MDS Clinical Research Consortium (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2014-0636
Record Dates: First submitted 2015-02-27; First posted 2015-03-04 (Estimated); Last update posted 2022-07-29 (Actual); Status verified 2022-07

CONDITIONS: Leukemia
Keywords: Leukemia; Myelodysplastic syndrome; MDS; Low- or intermediate-1-risk; Chronic Myelomonocytic Leukemia -1; CMML-1; Quality of Life in Myelodysplasia Scale; QUALMS-1; Anemia Subset of FACT; FACT-An; Questionnaires; Surveys
MeSH Terms: conditions — Leukemia; Myelodysplastic Syndromes | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Quality of Life in Myelodysplasia Scale (QUALMS-1): Participants complete the Quality of Life in Myelodysplasia Scale (QUALMS-1) and the Anemia Subset of FACT (FACT-An), instrument twice: at the start of treatment, and after four cycles or discontinuation of treatment, whichever comes first.
  Interventions: Behavioral: QUALMS-1 Questionnaire; Behavioral: FACT-An Questionnaire

INTERVENTIONS:
Behavioral: QUALMS-1 Questionnaire — Participants complete the QUALMS-1 during first treatment visit, and after 4th cycle of treatment or when treatment stops.
  Other Names: Survey
Behavioral: FACT-An Questionnaire — Participants complete the FACT-An during first treatment visit, and after 4th cycle of treatment or when treatment stops.
  Other Names: Survey

SUMMARY:
The goal of this research study is to test a quality-of-life questionnaire called QUALMS-1 in patients with MDS.

This is an investigational study.

Up to 240 participants will be enrolled in this multicenter study. Up to 175 will take part at MD Anderson.

DETAILED DESCRIPTION:
If you agree to take part in this study, you will be asked to complete questionnaires twice during your participation in the 2014-0112 study.

During your first treatment visit, you will be asked to complete the QUALMS-1 questionnaire and another questionnaire that asks about your well-being.

After your 4th cycle of treatment or when you stop receiving treatment, you will be asked to complete the QUALMS-1 questionnaire again and another questionnaire to rate any changes in your health since you started the study.

It should take about 20 minutes total to complete the questionnaires each time.

Information will also be collected from your medical record. This information will include the results of lab tests and other information relating to your health.

Length of Study Participation:

After you complete the questionnaires the second time, your participation in this study will be complete.

ELIGIBILITY:
Inclusion Criteria:

1. Sign an Institutional Review Board (IRB)-approved informed consent document.
2. Age greater than or equal to 18 years
3. de novo or secondary International Prognostic Scoring Status (IPSS) low- or intermediate-1-risk MDS, including Chronic Myelomonocytic Leukemia (CMML)-1
4. Eastern Cooperative Oncology Group (ECOG) performance status of greater than or equal to 3 at study entry
5. Organ function as defined below: Serum creatine greater than or equal to mg/dL x upper limit of normal (ULN); Total bilirubin greater than or equal to 2 x ULN; Alanine transaminase (ALT; Serum glutamic pyruvic transaminase=SGPT) greater than or equal to 2 x ULN
6. Women of childbearing potential must have a negative serum or urine pregnancy test within 7 days and will also need to use contraceptives. Men must agree not to father a child and agree to use a condom if his partner is of child bearing potential.

Exclusion Criteria:

1. Breast feeding females
2. Prior therapy with decitabine or azacitidine
3. Prior participation in the development of the QUALMS-1 (Dana-Farber Cancer Institute=DFCI)
4. Non-English speaking patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with myelodysplastic syndrome (MDS) taking part in the 2014-0112 study.
Sampling Method: Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2022-07-18 (Actual); Study Completion 2022-07-18 (Actual)

PRIMARY OUTCOMES:
Change in Quality of Life (QOL) | 4 months
  Participants rate any change in their quality of life since enrollment using a 7-point Likert-type change rating scale, ranging from much better, to no change, to much worse. This change rating scale used to characterize the QUALMS-1's reliability compared to its first administration as well as its responsiveness.

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Garcia-Manero, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (6):
- United States (6):
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - The Johns Hopkins University, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Weill Medical College of Cornell University, New York, New York
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - University of Texas MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org